CLINICAL TRIAL: NCT07292324
Title: Effectiveness of Continuous Epidural With Dexmedetomidine Adjuvant Compared to Without Adjuvant in Gynecologic Laparotomy
Brief Title: Continuous Epidural With Dexmedetomidine Adjuvant in Gynecologic Laparotomy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Simson Samuel Soerodjotanojo, Anesthesiology Resident, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2171102008
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Pain, Acute; Chronic Post Surgical Pain; Gynecologic Disease
Keywords: Dexmedetomidine; Bupivacaine; Epidural Analgesia; Gynecologic Laparotomy; NF-kappa B
MeSH Terms: conditions — Pain, Postoperative; Genital Diseases, Female | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P1 (Dexmedetomidine Adjuvant) (Experimental): Participants receive epidural analgesia with Bupivacaine 0.1% combined with Dexmedetomidine 0.5 mcg/ml. This is administered as a 10 ml loading dose before incision, followed by a continuous infusion (PCEA) at a rate of 3 ml/hour, with a demand dose of 5 ml and a lockout interval of 30 minutes for 24 hours post-operation.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- Group P2 (Control) (Active Comparator): Participants receive epidural analgesia with Bupivacaine 0.1% alone (without adjuvant). This is administered as a 10 ml loading dose before incision, followed by a continuous infusion (PCEA) at a rate of 3 ml/hour, with a demand dose of 5 ml and a lockout interval of 30 minutes for 24 hours post-operation.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine & Bupivacaine. — Epidural administration of Bupivacaine 0.1% combined with Dexmedetomidine 0.5 mcg/ml. Subjects receive a loading dose of 10 ml before incision. This is followed by a continuous infusion using Patient-Controlled Epidural Analgesia (PCEA) with a background rate of 3 ml/hour, a demand dose of 5 ml, and a lockout interval of 30 minutes for 24 hours post-operation.
  Arms: Group P1 (Dexmedetomidine Adjuvant)
Drug: Bupivacain — Epidural administration of Bupivacaine 0.1% without adjuvant. Subjects receive a loading dose of 10 ml before incision. This is followed by a continuous infusion using Patient-Controlled Epidural Analgesia (PCEA) with a background rate of 3 ml/hour, a demand dose of 5 ml, and a lockout interval of 30 minutes for 24 hours post-operation.
  Arms: Group P2 (Control)

SUMMARY:
The goal of this clinical trial is to learn if adding a medication called dexmedetomidine to an epidural block works better than a standard epidural to control pain in women undergoing gynecologic laparotomy (abdominal surgery). The main questions it aims to answer are:

Does adding dexmedetomidine reduce pain scores and the need for extra pain medicine in the first 24 hours after surgery? Does it lower inflammation levels and reduce the risk of developing chronic pain 3 months later?

Participants will receive an epidural (pain medicine delivered through a small tube in the back) combined with general anesthesia for their surgery. Researchers will compare two groups:

One group will receive the standard epidural medicine (bupivacaine) mixed with dexmedetomidine.

The other group will receive the standard epidural medicine (bupivacaine) alone.

Researchers will measure the participants' pain levels, how much pain medicine they use, and blood markers for inflammation for 24 hours after surgery. They will also contact participants 3 months later to check for any long-term pain.

DETAILED DESCRIPTION:
This is a double-blind, randomized, pre- and post-test control group study to evaluate the effectiveness of adding dexmedetomidine as an adjuvant to continuous epidural analgesia for patients undergoing gynecologic laparotomy.

Postoperative pain following laparotomy can be severe and is associated with inflammation and a risk of developing chronic postsurgical pain (CPSP). While epidural analgesia is a standard method for pain management, this study investigates whether the addition of dexmedetomidine (an alpha-2 adrenergic agonist) provides superior analgesia and anti-inflammatory effects compared to local anesthetic alone.

Participants aged 30-55 with ASA physical status I-III will be randomized into two groups:

Group P1 (Intervention): Receives an epidural bolus and continuous infusion of bupivacaine 0.1% combined with dexmedetomidine 0.5 mcg/ml.

Group P2 (Control): Receives an epidural bolus and continuous infusion of bupivacaine 0.1% alone.

The epidural catheter will be inserted at the L1-L2 level prior to the induction of general anesthesia. Postoperative pain will be managed using a Patient-Controlled Epidural Analgesia (PCEA) pump with specific settings (3 ml/hr background infusion, 5 ml bolus demand, 30-minute lockout).

Key outcome measures include:

Acute Pain: Visual Analogue Scale (VAS) scores recorded at 6, 12, and 24 hours post-operation.

Analgesic Consumption: Total volume of bupivacaine used and total PCEA demands in 24 hours.

Inflammatory Response: Changes in Nuclear Factor Kappa B (NFκB) levels measured from blood samples taken pre-operatively and 24 hours post-operatively.

Chronic Pain: Incidence of chronic pain assessed 3 months post-operatively using the Brief Pain Inventory Short Form (BPI-SF).

Safety: Monitoring for adverse events such as hypotension and bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-55 years
* ASA physical status I-III
* Body Mass Index (BMI) 18 - 29.9 kg/m2
* Patients undergoing gynecologic laparotomy

Exclusion Criteria:

* Contraindications for regional anesthesia
* Allergy or contraindication to dexmedetomidine
* Routine use of antidepressants or anticonvulsants
* Chronic opioid consumption (equivalent to >30 mg oral morphine per day for >1 month)
* History of Chemotherapy-Induced Peripheral Neuropathy (CIPN)
* Active systemic autoimmune disease or receiving immunosuppressant therapy (e.g., Systemic Lupus Erythematosus, Rheumatoid Arthritis, Multiple Sclerosis)
* Inability to use the Visual Analogue Scale (VAS) or operate the Patient-Controlled Epidural Analgesia (PCEA) device
* Coagulation disorders (prolonged hemostasis)
* Refusal to participate

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (VAS) | 6, 12, and 24 hours post-operation
  Pain intensity is assessed using the Visual Analogue Scale (VAS). The VAS consists of a 100 mm straight line where the left end indicates "no pain" and the right end indicates "very severe pain" (0-100 mm). Participants mark the line to indicate their pain level. Higher scores indicate worse pain

SECONDARY OUTCOMES:
Total Bupivacaine Consumption | 24 hours post-operation.
  The total volume of Bupivacaine (in milliliters) consumed via the Patient-Controlled Epidural Analgesia (PCEA) pump during the postoperative period.
Total PCEA Demands | 24 hours post-operation.
  The total number of times the participant pressed the PCEA button to request an analgesic bolus dose (total demand).
Change in Nuclear Factor Kappa B (NFκB) Level | Baseline (Pre-operative) and 24 hours post-operation.
  The difference in serum levels of the inflammatory biomarker Nuclear Factor Kappa B (NFκB). This is calculated as the value at 24 hours post-operation minus the pre-operative baseline value.
Incidence of Chronic Postsurgical Pain | 3 months post-operation.
  The occurrence of chronic pain assessed using the Brief Pain Inventory Short Form (BPI-SF). The BPI-SF measures pain severity (worst, least, average, now) and pain interference with daily activities. Scores range from 0 to 10, with higher scores indicating worse pain/interference .
Incidence of Bradycardia | Up to 24 hours post-operation.
  The number of participants experiencing bradycardia, defined as a heart rate less than 50 beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Simson Samuel Soerodjotanojo, Principal Investigator — Udayana University; I Gusti Ngurah Mahaalit Aribawa, Study Director — Udayana University; I Made Agus Kresna Sucandra, Study Director — Udayana University
Locations (1):
- Prof. Dr. I.G.N.G Ngoerah Central General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao Y, Chen Z, Huang Y, Sun S, Yang D. Comparison of dexmedetomidine and opioids as local anesthetic adjuvants in patient controlled epidural analgesia: a meta-analysis. Korean J Anesthesiol. 2024 Feb;77(1):139-155. doi: 10.4097/kja.22730. Epub 2023 May 2. PMID 37127531
- [Background] Zhang X, Wang D, Shi M, Luo Y. Efficacy and Safety of Dexmedetomidine as an Adjuvant in Epidural Analgesia and Anesthesia: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Clin Drug Investig. 2017 Apr;37(4):343-354. doi: 10.1007/s40261-016-0477-9. PMID 27812971
- [Background] Hetta DF, Fares KM, Abedalmohsen AM, Abdel-Wahab AH, Elfadl GMA, Ali WN. Epidural dexmedetomidine infusion for perioperative analgesia in patients undergoing abdominal cancer surgery: randomized trial. J Pain Res. 2018 Oct 30;11:2675-2685. doi: 10.2147/JPR.S163975. eCollection 2018. PMID 30464585